CLINICAL TRIAL: NCT03002961
Title: A Multicenter, Open-Label, Single Ascending-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Depot Buprenorphine (RBP-6000) in Opioid-Dependent Subjects
Brief Title: Single Ascending Dose Study of RBP-6000
Acronym: SAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-11-0020
Record Dates: First submitted 2016-12-15; First posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): Subjects to receive low dose of RBP-6000 subcutaneously as a single injection
  Interventions: Drug: RBP-6000
- Cohort 2 (Experimental): Subjects to receive medium dose of RBP-6000 subcutaneously as a single injection
  Interventions: Drug: RBP-6000
- Cohort 3 (Experimental): Subjects to receive high dose of RBP-6000 subcutaneously as a single injection
  Interventions: Drug: RBP-6000
- Cohort 4 (Experimental): Subjects would receive medium dose RBP-6000 as a single injection after up to 12 mg daily dosing of sublingual (SL) suboxone tablets for 7 days
  Interventions: Drug: RBP-6000; Drug: Suboxone

INTERVENTIONS:
Drug: RBP-6000 — single dose of RBP-6000, preceded by a pharmacokinetic (PK) sample followed by serial PK samples post-dose. Additionally subjects to remain in the clinic through Day 21 for safety assessments
  Other Names: atrigel buprenorphine
Drug: Suboxone — RBP-6000 injection after 7 days of SL Suboxone administration. Interventions as above with additional daily PK collections during Suboxone treatment prior to RBP-6000 administration
  Arms: Cohort 4

SUMMARY:
A multi-center, open-label, single ascending dose study to enroll opioid dependent treatment-seeking subjects. Subjects to be enrolled into 3 cohorts receiving low, medium and high doses of depot buprenorphine. A fourth cohort will be enrolled to evaluate the PK of RBP-6000 after receiving suboxone tablets for 7 days.

DETAILED DESCRIPTION:
All subjects will undergo screening period of up to 7 days. Eligible subjects in Cohorts 1-3 will receive RBP-6000 doses on at the conclusion of screening. Subjects in Cohort 4 will receive sublingual (SL) Suboxone for 7 days prior to receiving an injection of RBP-6000.

For all cohorts, subjects will be admitted to the clinic 2 days prior to beginning any dosing, and will remain in the clinic through Day 21. Blood collection for hematology, chemistry and serology analysis will be drawn at screening, and intermittently for safety assessments during the study period. Subjects in Cohorts 1-3 will have a PK sample collected pre-dose and serial PK collection post-dosing. Subjects in Cohort 4 will have daily PK collections while admitted during Suboxone dosing and serially after RBP-6000 administration.

Subjects will return to the clinic for PK sample collection through Day 140 or until buprenorphine concentrations fall below 100 pg/mL. Subjects will return to the clinic for safety assessments through Day 150.

Subjects experiencing signs and symptoms of withdrawal prior to RBP-6000 during the residential phase may receive non-opioid rescue medications. Subjects who experience signs and symptoms of withdrawal may receive hydromorphone beginning on Day 11 if necessary. Methadone dosing can begin, if clinically indicated, on Day 16 only for subjects who have not been administered hydromorphone. Subjects will not be allowed to use buprenorphine at any time during the study.

Subjects will also receive psychosocial and behavioral counseling as specified by the PI. The End of Study visit will occur 1 week after Day 84 or 1 week after the monthly follow-up visits after Day 84, given a subject's buprenorphine plasma concentration has fallen below 100 pg/mL. For subjects with plasma concentrations of buprenorphine above 100 pg/mL at Day 140, Day 150 will be the End of Study visit.

Subjects will not be enrolled into the next cohort until safety data for at least the first 6 subjects has been reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male and female subjects are eligible for entry.
* Age: ≥ 18 to ≤ 65 years.
* Body mass index (BMI) of ≥ 18.0 to ≤ 33.0 kg/m2
* Female subjects must have a negative pregnancy test. Women of child bearing potential should have been surgically sterile for at least 6 months prior to dosing or must agree to take reasonable precautions during the study to avoid pregnancy by agreeing to remain abstinent or to practice one of the following methods of birth control from study screening through the last study visit: double barrier (e.g., diaphragm with spermicide; condoms with spermicide); intrauterine device (IUD); implanted or intrauterine hormonal contraceptives in use for at least 6 consecutive months prior to study dosing; or oral, patch, or injected contraceptives or vaginal hormonal device in use for at least 3 consecutive months prior to study.
* Meet DSM-IV-TR criteria for opioid dependence and are seeking opioid-dependence treatment.

(Note: Subjects need not to be seeking treatment with methadone but be willing to accept methadone treatment as consequence of the study.)

* Normal or no clinically significant electrocardiogram (ECG) findings at screening or through predose on Day 1.
* Total bilirubin ≤ 2x the upper limit of normal (ULN), alanine aminotransferase (ALT) ≤ 2xULN, aspartate aminotransferase (AST) ≤ 2xULN, serum creatinine ≤ 2xULN, and international normalized ratio (INR) ≤ 2xULN.
* Agree not to take any buprenorphine products other than those administered for the current study (SUBOXONE SL tablets and RBP-6000) throughout participation in the study.
* Willing to cooperate with study procedures and provide written informed consent prior to start of any study procedures.

Exclusion Criteria:

* Require ongoing opioid therapy for pain or other chronic medical conditions.
* ECG demonstrating QTc > 450 msec in males and QTc > 470 msec in females at clinic entry or prior to administration of RBP-6000.
* Currently dependent by DSM-IV-TR criteria on any substances other than opioids, caffeine, or nicotine.
* Currently (during past 30 days from the signing of the informed consent document) engaged in opioid agonist, partial agonist, or antagonist treatment; or require on-going prescription or over the counter (OTC) medications that are clinically relevant CYP P450 3A4 inducers or inhibitors (e.g., rifampicin, azole antifungals [e.g., ketoconazole], macrolide antibiotics [e.g., erythromycin]). See Appendix 12 for an excluded medications list.
* Significant traumatic injury, major surgery, or open biopsy within the prior 4 weeks of informed consent.
* Buprenorphine use within 30 days of informed consent.
* Subjects with a COWS score of < 12 on the day of administration of RBP-6000 (Applicable for subjects in Cohort 1-3 only, subjects for cohort 4 will not be excluded with a COWS score <12).
* Subjects with any history of suicidal ideation within 30 days prior to informed consent or study drug administration as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the C-SSRS completed at the screening visit, or any history of suicide attempts.
* Clinically significant abnormality in past medical history or at the screening physical examination that in the opinion of the PI or Sponsor may place the volunteer at risk or interfere with outcome variables including absorption, distribution, metabolism, and excretion of drug, including but is not limited to history or concurrent cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease.
* History or presence of allergic or adverse response (including rash or anaphylaxis) to buprenorphine, naloxone, methadone, or the ATRIGEL Delivery System.
* Donation of> 250 mL of blood or plasma or participation in another clinical trial within 30 days prior to signing of the informed consent document for this study.
* Current use of or positive urine screen at clinic admission for barbiturates, benzodiazepines, buprenorphine, or methadone.
* Serology positive for human immunodeficiency virus (HIV), acute hepatitis B, or acute hepatitis C and subjects positive for both hepatitis B surface antigen (HBsAg) and immunoglobulin M antibodies to hepatitis B core antigen (anti-HBc IgM). (Note: Subjects with asymptomatic hepatitis B or C infection may be enrolled.)
* All herbal supplements, grapefruit and grapefruit juices, and OTC medications. Sponsor may allow exceptions of medicines that are unlikely to impact PK or PD results.
* Subjects who have been previously excluded from participation or previously enrolled into the study or have previously participated in a study with RBP-6000.
* Subjects who are unable, in the opinion of the PI or the medically responsible physician, to comply fully with the study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety will be assessed by the frequency of adverse events (AEs), serious AEs, and discontinuations due to AEs (safety and tolerability) in subjects receiving a single dose of RBP-6000. | Baseline (defined as last non-missing value prior to dosing) to end of study/day 150 or early termination
  Safety will be assessed by AEs, ECGs, laboratory measurements, local injection site tolerability and vital signs
Individual, mean and median PK concentrations over time profiles will be plotted for subjects receiving a single dose of RBP-6000 with an adequate number of PK samples collected to derive PK parameters. | PK prior to injection through Day 150/End of Study or Early Termination
  Individual plasma concentrations will be collected to compute PK parameters. The individual concentrations will be summarized using descriptive statistics.
The safety of RBP-6000 when administered as a single SC injection after daily dosing of SL Suboxone will be assessed as a measure of the occurrence of AEs, serious AEs and discontinuations due to AEs | Day -7 through Day 150/End of Study or Early Termination
  Safety to be assessed by AEs, ECGs, laboratory measurements, local injection site tolerability and vital signs

SECONDARY OUTCOMES:
Change from baseline of subject suicidal ideation will be reported using the Columbia Suicide Severity Rating Scale (C-SSRS) | Screening through Day 150/End of Study or Early Termination
  Suicidal ideation scores will be reported using the Columbia Suicide Severity Rating Scale (C-SSRS).
Change from baseline of physician reported withdrawal symptoms will be reported by Clinical Opiate Withdrawal Scale (COWS) score | Screening through Day 150/End of Study or Early Termination
  Opioid withdrawal symptoms will be measured by Clinical Opiate Withdrawal Scale (COWS) score.
Change from baseline of subject reported withdrawal symptoms will be reported by Visual Analog Scale (VAS) total score | Screening through Day 150/End of Study or Early Termination
  Opioid withdrawal symptoms will be measured by Visual Analog Scale (VAS) total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Vince and Associates Clinical Research, Overland Park, Kansas, United States